CLINICAL TRIAL: NCT05412797
Title: Use of a DeskCycle to Reduce Sedentary Behavior During the Workday
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: DeskCycle (Unknown)
Responsible Party: Principal Investigator, Melissa Zullo, Professor of Epidemiology, Kent State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 17-226
Record Dates: First submitted 2022-05-04; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Chronic Disease; Reduction, Weight
MeSH Terms: conditions — Chronic Disease; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycling (Experimental): Used a DeskCycle during the workday/the intervention increased the amount of time spent being physically active.
  Interventions: Behavioral: Cycling/Using a DeskCycle
- Control (Active Comparator): Regular activities
  Interventions: Behavioral: Regular activities

INTERVENTIONS:
Behavioral: Cycling/Using a DeskCycle — The intervention was conducted in two phases. In phase 1, the intervention group were given the DeskCycles to use for 8 weeks. In phase, the control group from phase 1 were given the DeskCycles to use. Intervention group from phase 1 became controls in phase 2
  Arms: Cycling
Behavioral: Regular activities — The active comparator performed normal daily activities
  Arms: Control

SUMMARY:
The purpose of this research was to evaluate the effectiveness of a DeskCycle intervention in reducing sedentary behavior by increasing the time spent participating in light to moderate physical activity in a randomly selected group of desk job employees at Kent State University main campus. The study also assessed the feasibility of using the DeskCycle in the working environment, as well as the effect on weight and mood. The primary outcome of interest was the 'mean minutes of light to moderate physical activity'. Secondary outcomes include weight, mood score, and feasibility of using the DeskCycle. The study was a randomized controlled trial (RCT) with a cross-over design where differences between the intervention and control group were evaluated over an eight-week period, after which there was a switch and the DeskCycles were given to the control group to use for the eight-week period that followed. The allocation during the first eight-week period intervention will be done through random process.

ELIGIBILITY:
Inclusion Criteria:

* females 18 years and above
* full-time Kent State university administrative employees at the Kent main campus
* sedentary for 75% of their workday
* height under 5'10"
* desk height of at least 27"

Exclusion Criteria:

* any uncontrolled cardiovascular diseases
* back, knee or other joint pains

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-05-06 (Actual)

PRIMARY OUTCOMES:
Minutes of Exercise | Daily (M-F) for 8 weeks time period 1 and 2
  Mean minutes of light to moderate physical activity
Feasibility of using the deskcycle during work | Week 2 period 1 and 2
  How feasible was it to use the DeskCycle during work
Feasibility of using the deskcycle during work | Week 8 period 1 and 2
  How feasible was it to use the DeskCycle during work
Mood | Baseline period 1 and 2
  How was mood impacted during the work day
Mood | Week 4 period 1 and 2
  How was mood impacted during the work day
Mood | Week 8 period 1 and 2
  How was mood impacted during the work day

SECONDARY OUTCOMES:
Change in weight | Baseline to end of study period 1 and 2
  Bodyweight before and after the study

CONTACTS AND LOCATIONS:
Locations (1):
- Kent State University, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No